CLINICAL TRIAL: NCT03822403
Title: Randomized, Controlled Clinical Evaluation of Glass Ionomer System vs Composite Posterior Restorations
Brief Title: Clinical Performance Evaluation of a Glass-ionomer Restorative System Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEK 09/112-11
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Dental Caries
Keywords: glass ionomer; composite resin
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EQUIA (Active Comparator): EQUIA Placing glass ionomer restorations, the dentin and enamel of cavities were conditioned with 20% polyacrylic acid for 20 seconds, washed, and briefly dried. Equia Fil was injected into the cavity. Isolation was maintained using cotton rolls and a saliva ejector. After the setting time of 2.5 minutes, the restoration was polished wet using high-speed fine diamonds. When the restoration was briefly dried, Equia Coat was applied and photocured for 20 seconds using a photo-curing light.
  Interventions: Device: EQUIA
- Gradia Direct Posterior (Active Comparator): Gradia Direct Posterior The enamel and dentin were conditioned with G-Bond adhesive using a microtip applicator, left undisturbed for five to 10 seconds, and then dried thoroughly for five seconds with oil-free air under air pressure, Gradia Direct Posterior resin was applied with the incremental technique (2 mm thick layers) and light-cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments.
  Interventions: Device: Gradia Direct Posterior

INTERVENTIONS:
Device: EQUIA — Placing glass ionomer restorations, the dentin and enamel of cavities were conditioned with 20% polyacrylic acid for 20 seconds, washed, and briefly dried. Equia Fil was injected into the cavity. Isolation was maintained using cotton rolls and a saliva ejector. After the setting time of 2.5 minutes, the restoration was polished wet using high-speed fine diamonds. When the restoration was briefly dried, Equia Coat was applied and photocured for 20 seconds using a photo-curing light.
  Other Names: Glass ionomer restorative system
  Arms: EQUIA
Device: Gradia Direct Posterior — The enamel and dentin were conditioned with G-Bond adhesive using a microtip applicator, left undisturbed for five to 10 seconds, and then dried thoroughly for five seconds with oil-free air under air pressure, Gradia Direct Posterior resin was applied with the incremental technique (2 mm thick layers) and light-cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments.
  Other Names: Micro hybrid composite
  Arms: Gradia Direct Posterior

SUMMARY:
The aim of this clinical trial was to compare the clinical performances of a glass ionomer restorative system with a micro hybrid resin based composite in class I and class II cavities. A total of 140 (80 class I and 60 class II) lesions in 59 patients were restored with a glass ionomer restorative system (Equia) or a micro hybrid composite(Gradia Direct). Restorations were evaluated at baseline and yearly during 9 years according to the modified-USPHS criteria. Data were analyzed with Cohcran's Q and McNemar's tests (p<0.05).

DETAILED DESCRIPTION:
Since the introduction of glass ionomers many modifications of these materials have been performed over the years. Compared to other permanent filling materials like resin-based composites, glass ionomers show several advantages, such as the ability to adhere to moist enamel and dentin and anti- cariogenic properties such as the long-term fluoride release. So, it was doubtful that glass ionomers represent a capable counterpart of amalgam or resin-based composites in posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

1. a need for at least two but not more than four posterior toothcolored restorations;
2. the presence of teeth to be restored in occlusion;
3. teeth that were symptomless and vital;
4. a normal periodontal status;
5. a good likelihood of recall availability.

Exclusion Criteria:

1. partly erupted teeth;
2. absence of adjacent and antagonist teeth
3. poor periodontal status;
4. adverse medical history;
5. potential behavioral problems.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria Observers evaluated the restorations was performed using the modified United State Public Health Service criteria Marginal adaptation | From baseline to 9 year the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap (max 100μ) with discoloration (removable)
marginal discoloration | From baseline to 9 year the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal discoloration. Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth. Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction
retention rate | From baseline to 9 year the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed .
  A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
anatomic form | From baseline to 9 year the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding anatomic form. Anatomic form was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed .
  A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture.
color change | From baseline to 9 year the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding color change. Colour changes was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: The restoration matches the adjacent tooth structure in color and translucency.
  Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University School of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gurgan S, Kutuk ZB, Ergin E, Oztas SS, Cakir FY. Four-year randomized clinical trial to evaluate the clinical performance of a glass ionomer restorative system. Oper Dent. 2015 Mar-Apr;40(2):134-43. doi: 10.2341/13-239-C. Epub 2014 Oct 9. PMID 25299703
- [Background] Gurgan S, Kutuk ZB, Ergin E, Oztas SS, Cakir FY. Clinical performance of a glass ionomer restorative system: a 6-year evaluation. Clin Oral Investig. 2017 Sep;21(7):2335-2343. doi: 10.1007/s00784-016-2028-4. Epub 2016 Dec 20. PMID 28000039
- [Background] Turkun LS, Kanik O. A Prospective Six-Year Clinical Study Evaluating Reinforced Glass Ionomer Cements with Resin Coating on Posterior Teeth: Quo Vadis? Oper Dent. 2016 Nov/Dec;41(6):587-598. doi: 10.2341/15-331-C. Epub 2016 Aug 29. PMID 27571238